CLINICAL TRIAL: NCT01906203
Title: Evaluation of Indices of Body Composition During Ultramarathon : Measure by Body Bioelectrical Impedance
Acronym: IMPETRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0163
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
Keywords: Ultramarathon; bioelectrical impedance; Phase-Angle

ARMS (1):
- ultramarathon (Experimental)
  Interventions: Device: body bioelectrical impedance performed by Z-Métrix (class IIa) - BIOPARHOM 12 allée des lacs de garde, Savoie Technolac BP 238, 73374 Bourget du lac, France

INTERVENTIONS:
Device: body bioelectrical impedance performed by Z-Métrix (class IIa) - BIOPARHOM 12 allée des lacs de garde, Savoie Technolac BP 238, 73374 Bourget du lac, France

SUMMARY:
Prospective cohort, monocentric non-randomized and interventional clinical study in ICU assessing the evolution of body composition using bioelectrical impedance analysis.

DETAILED DESCRIPTION:
Prospective, monocentric non-randomized and interventional clinical study in ICU assessing the evolution of body composition using bioelectrical impedance analysis (phase angle, fat mass, muscle mass, fat-free mass, body water) before and after ultramarathon.

ELIGIBILITY:
Inclusion Criteria:

* Participation to ultramarathon

Exclusion Criteria:

* pregnancy women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Difference of fat-free mass, using bioelectrical impedance analysis | before and after ultramarathon of 105 km (at day 1)

SECONDARY OUTCOMES:
Difference of phase angle, using bioelectrical impedance analysis | at day 1(before and after ultramarathon)
Correlation between order in the course,duration of course and indices of body composition | at day 1 (during ultramarathon of 105 km)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France